CLINICAL TRIAL: NCT01169181
Title: AMES + Brain Stimulation: Treatment for Profound Plegia in Stroke
Brief Title: AMES + Brain Stimulation
Acronym: AMES
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AMES Technology (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6237; 1R43NS067694-01A1 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Stroke; Cerebrovascular Accident; Plegia
Keywords: Stroke; Cerebrovascular Accident; Plegia; Upper Extremity; rTMS; tDCS
MeSH Terms: conditions — Stroke; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMES therapy with rTMS (Active Comparator): Each subject will participate in 30 therapy sessions over a 10- to 15-week period. A session will last 90 to 120 minutes, which includes 20 minutes of AMES+rTMS, followed by an EMG test. During the hand-opening phase of the AMES therapy, the subjects assigned to the AMES+rTMS treatment group will be subjected to trains of TMS pulses.
  Interventions: Device: AMES + brain stimulation
- AMES therapy with tDCS (Active Comparator): Each subject will participate in 30 therapy sessions over a 10- to 15-week period. A session will last 90 to 120 minutes, which includes 20 minutes of AMES+tDCS, followed by an EMG test. A constant current will be applied throughout the entire 20-minute therapy session with the AMES device.
  Interventions: Device: AMES + brain stimulation

INTERVENTIONS:
Device: AMES + brain stimulation — Stroke survivors with plegia of affected upper extremity receive either AMES + rTMS or AMES + tDCS.

SUMMARY:
The procedure involves: (1) assisted hand movement by a mechanical device, (2) mechanical vibration applied to the surface of the forearm, and (3) stimulation of the brain with either transcranial magnetic stimulation (TMS) or transcortical direct current stimulation (DCS). These 3 components of the procedure are carried out simultaneously. Each subject will be evaluated pre- and post-treatment with several clinical tests of functional movement. The hypotheses of this project are that the AMES+rTMS and AMES+tDCS procedures are safe and will enable most of the stroke patients to recover finger extension.

DETAILED DESCRIPTION:
This protocol is designed to investigate the safety and efficacy of a procedure for treating chronic (>1 year post) stroke patients who still cannot move the hand affected by the stroke. The treatment involves: (1) assisted hand movement by a mechanical device, (2) mechanical vibration applied to the surface of the forearm, and (3) stimulation of the brain with either transcranial magnetic stimulation (TMS) or transcortical direct current stimulation (DCS). Subjects receiving TMS during treatment are expected to respond more fully (i.e., increased volitional EMG) in the treated hand compared to those receiving DCS.

ELIGIBILITY:
Inclusion Criteria:

* Stroke occurring ≥12 months before enrollment
* Hemispheric stroke (ischemic or hemorrhagic), cortical or subcortical
* Residual upper-extremity weakness without the ability to activate volitionally extensor digitorum (no volitional EMG in the long finger extensor muscle)independently
* Age 18-75 years old

Exclusion Criteria:

* Significant upper-extremity proprioceptive deficit (<70% correct detection of the direction of passive finger movement, with eyes closed)
* Cortical stroke involving the primary motor cortex
* Epilepsy not controlled by medication
* Botox injections 5 months before or during enrollment; use of intrathecal Baclofen
* Residual pain in the tested arm
* Significant neglect involving the affected limb (NIHSS 2 on the extinction and attention items)
* Exercise intolerant
* Uncontrolled hypertension or angina
* Cognitive or behavioral inability to follow instructions
* Current abuse of alcohol or drugs
* Terminal illness with anticipated survival of <12 months
* Severe apraxia; inability to understand oral directions in English; or inability to communicate adequately with study personnel
* Circumference of arm incompatible with the AMES device (checked by placing the limb in the device)
* Contractures, decreased range of motion, or skin condition preventing tolerance of the AMES muscle vibrators
* Spinal cord injury, arthritis, or fractures of affected limbs resulting in loss of range of motion
* In the tested arm, peripheral nerve injury or neuropathy resulting in significant motor or sensory loss
* Pathological neurological/physical condition other than stroke that impairs the function of the impaired arm or that produces pain in the impaired arm
* Implanted device (e.g., cardiac pacemaker, Baclofen pump) the operation of which might be adversely affected by the brain stimulation
* Previous vascular surgery on the blood vessels of the brain or heart or heart valve surgery
* Female and pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maximum volitional EMG in the extensor digitorum and the finger flexors | Following each treatment with the AMES device
  EMG intensity will be measured during maximal efforts at hand opening and closing at the end of each treatment session. The averages of 3 attempted openings and 3 closings will be determined and recorded.

SECONDARY OUTCOMES:
Chedoke-McMaster Stroke Assessment | Before the first treatment session, and again after the last treatment session.
  A validated assessment tool for evaluating the severity of physical impairment in adult stroke survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University; Paul J. Cordo, PHD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411